CLINICAL TRIAL: NCT03406572
Title: Comparison of High Flow Nasal Cannula Oxygen and Conventional Oxygen Therapy on Ventilatory Support Duration During Acute-on-chronic Respiratory Failure: a Multicenter, Randomized, Controlled Trial
Brief Title: Use of Nasal High Flow Oxygen During Breaks of Non-invasive Ventilation for Patients With Hypercapnic Respiratory Failure
Acronym: HIGH FLOW ACRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Direction Générale de l'Offre de Soins (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: K160911J
Record Dates: First submitted 2017-11-23; First posted 2018-01-23 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Hypercapnic Respiratory Failure
Keywords: Acute on chronic respiratory failure; High-Flow heated and humidified nasal oxygen therapy
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFHO Group (Experimental): Patients will receive a first NIV session (for 2 hours) with predefined parameters, and ABG will be performed between one and two hours of starting NIV. NIV will be extended according to ABG result (i.e. extended if pH < 7.30). Switch from NIV to oxygen will require predefined criteria. In-between each NIV session, oxygen will be delivered using a high flow nasal cannula, with a flow of 50-60L/min and a FiO2 set to reach a targeted SpO2: 88%≤SpO2 ≤ 92%. Predefined criteria will be used to resume NIV.
  Interventions: Device: HFHO Group
- Standard O2 Group (Active Comparator): NIV will be initiated based on the same criteria and with the same parameters as the HFHO group. ABG will also be performed between one and two hours and NIV extended according to ABG result (i.e. extended if pH < 7.30). Switch from NIV to oxygen will require the same predefined criteria as the HFHO group. In-between each NIV session, oxygen will be delivered using standard low flow O2 to reach the same targeted SpO2: 88% ≤SpO2 ≤ 92%. Similar criteria will be used to resume NIV
  Interventions: Device: Standard O2

INTERVENTIONS:
Device: HFHO Group — * Common name: humidifier with integrated flow generator that delivers high flow warmed and humidified respiratory gases
  * Brand name: Airvo 2
  Other Names: High-flow heated and humidified nasal oxygen therapy (HFHO).
  Arms: HFHO Group
Device: Standard O2 — Standard oxygen therapy
  Arms: Standard O2 Group

SUMMARY:
Chronic respiratory insufficiency and COPD are the third leading cause of death worldwide. Patients decompensate at various stages of their disease and exhibit acute-on-chronic respiratory failure (ACRF), a frequent cause of ICU hospitalization for hypercapnic acute respiratory failure (ARF). Non-invasive ventilation (NIV) is the first line ventilatory treatment for hypercapnic ARF. It is applied intermittently, separated by periods of spontaneous breathing (SB) with standard oxygen (O2).

Standard O2 has drawbacks that limit the benefit of intermittent NIV in hypercapnic ARF: limited gas flow which is well below the patient's inspiratory flow rate, limited capacity and efficiency of oxygenation with non-controlled FiO2 (risk of excessive oxygen and induced hypercapnia), and cold and dry gas leading to discomfort and under-humidification of the airways and tracheobronchial secretions. Benefits in terms of work of breathing and CO2 removal resulting from PEEP and pressure support applied during NIV periods could be rapidly lost during standard O2.

Recently, use of high-flow heated and humidified nasal oxygen therapy (HFHO) has gained enthusiasm among intensivists to manage ARF. HFHO delivers high flows (up to 60L/min, that generate moderate PEEP) of heated and humidified oxygen at a controlled and adjustable FiO2 (21 to 100%) that rapidly improve respiratory distress symptoms, oxygenation, respiratory comfort and outcome of patients with hypoxemic ARF.

These unique features of HFHO could overcome some of the drawbacks of standard O2 during SB periods in hypercapnic ARF. Indeed, PEEP effect, washout of nasopharyngeal dead-space limiting CO2 re-breathing and inspired gas conditioning preserving adequate mucosal function and secretion removal, could potentially contribute to decrease airways resistance, intrinsic PEEP and work of breathing, while improving patient comfort. Investigators aim to determine if the use of HFHO, as compared to standard O2, increases the number of ventilator-free days (VFDs) and alive at day 28 in patients with hypercapnic ARF admitted in an ICU, an intermediate care, or a respiratory care unit, and requiring NIV.

DETAILED DESCRIPTION:
In both groups, treatment will start with a first NIV session of 2 hours, with arterial blood gas measurement between one hour and two hours after initiating the NIV session. The NIV will be extended for those patients with a pH < 7.30. In both groups, patients will be assessed for their tolerance of NIV and their ability to switch to spontaneous breathing every hour +/- 30 min, except during sleep (10 pm-8 am); they will be assessed for their tolerance of spontaneous breathing and for the need of resumption of NIV every 2 hours+/- 30 min and every 4 +/- 1 hours thereafter. To ensure the consistency of indications of NIV and invasive mechanical ventilation (IMV) across centers and reduce potential bias, NIV and IMV will be initiated and stopped in the same way in the two groups, using predefined criteria.

* Inclusion (day 0): informed consent, randomisation (HFHO group/standard O2 group), NIV initiation (for 2 hours), clinical and paraclinical exam including ABG, data collection
* Follow-up (day 1 to day 28) : NIV, clinical exam, ABG, data collection

ELIGIBILITY:
Inclusion criteria

* Adult patients aged 18 or above, admitted to an ICU, an intermediate care or a respiratory care unit;
* Chronic respiratory disease previously documented or strongly suspected on clinical, radiological and blood gazes data and pulmonary function tests, in connection with an obstructive respiratory disease (COPD, emphysema, overlap-syndrome (COPD + obstructive sleep apnoea) or mixed (bronchiectasis, obesity-hypoventilation syndrome))
* Patients requiring NIV for hypercapnic ARF (whatever the precipitating cause) i.e. with clinical signs of moderate to severe respiratory distress : dyspnea and /or respiratory rate > 25/min and/or use of accessory respiratory muscles and/or paradoxical abdominal motion and/or signs of respiratory encephalopathy (sleepiness, asterixis, confusion); and respiratory acidosis on arterial blood gases, defined by pH<7.35 and PaCO2 > 45 mmHg despite the careful supply of oxygen and appropriate therapy that may include bronchodilators, corticosteroids and antibiotics

Exclusion criteria

* Contraindications to NIV;
* Purely restrictive lung disease (thoracic deformity, neuro-muscular pathology) and pure obstructive sleep apnoea (without spirometric disturbance or daytime gas anomaly)
* Immediate need for intubation (respiratory or cardiac arrest);
* Persistent hemodynamic instability (use of vasopressors for > 1 hour);
* Multiple organ failure (score SOFA>6);
* NIV treatement for >3 consecutive hours (without any interruption) before admission to ICU, intermediate care, or respiratory care unit and before randomization;
* Anticipated difficulties to conduct NIV (facial trauma or deformation, edentulous patient);
* End stage chronic respiratory insufficiency (defined as use of NIV at home or CPAP treatment at home and life expectancy below 6 month);
* Non-treated pneumothorax;
* Impossibility to perform subjective assessment of dyspnea and comfort (cognitive impairment);
* Patient under guardianship or trusteeship;
* Pregnancy/breastfeeding;
* Decision to withhold or to withdraw life-sustaining treatments (including intubation)
* Moribund state
* Current participation in another clinical trial with an endpoint related to NIV.
* No affiliation to social security (beneficial or assignee);
* Refusal to participate to the study (patient or legal representative or family member or close relative if present

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2023-06-18 (Actual); Study Completion 2023-08-18 (Actual)

PRIMARY OUTCOMES:
Number of ventilator-free days (VFDs) alive | At day 28 after study enrollment

SECONDARY OUTCOMES:
Delay of completion of stopping rules for NIV | 28 days post-randomisation
Patient self-assessement of comfort during each SB period measured by Visual Analog Scale (score range 0-10, higher values represent a better outcome) | After 2 hours of SB in the 48 first hours, and every 4 hours thereafter, up to 28 days
Nurse assessement of comfort during each SB period measured by Likert scale (score range1-5; higher values represent a better outcome) | After 2 hours of SB in the 48 first hours, and every 4 hours thereafter, up to 28 days
Hospital length of stay | 28 days post-randomisation
All cause mortality | 28 days post-randomisation
Proportion of patients with facial skin erythema and/or ulceration | After 2 hours of SB in the 48 first hours, and every 4 hours thereafter; and after 1 hour of NIV; up to 28 days
Number of NIV sessions | 28 days post-randomisation
Duration of NIV sessions (hours) | 28 days post-randomisation
Number of days between the day the patient first meets criteria for NIV cessation and day 28 post-randomization | 28 days post-randomisation
Number of days between the day of initially achieving unassisted ventilation and day 28 post-randomization (i.e. after having successfully spent 48 consecutive hours of unassisted breathing) | 28 days post-randomisation
Proportion of patients achieving 48 consecutive hours of daytime unassisted breathing | 28 days post-randomisation
Proportion of patients requiring NIV resumption after 48 consecutive hours of daytime unassisted breathing | 28 days post-randomisation
Patient self-assessement of comfort during each NIV period measured by Visual Analog Scale (score range 0-10, higher values represent a better outcome) | after 1 hour of NIV, up to 28 days
Nurse assessement of comfort during each NIV period measured by Likert scale (score range1-5; higher values represent a better outcome) | after 1 hour of NIV, up to 28 days
Patient self-assessement of dyspnea during each SB period measured by Visual Analog Scale (range 0-10; higher values represent a worst outcome) | after 2 hours of SB in the 48 first hours, and every 4 hours thereafter, up to 28 days
Nurse assessement of dyspnea during each SB period measured by Likert scale (score range1-5; higher values represent a worst outcome) | after 2 hours of SB in the 48 first hours, and every 4 hours thereafter, up to 28 days
Patient self-assessement of dyspnea during each NIV period measured by Visual Analog Scale (range 0-10; higher values represent a worst outcome) | after 1 hour of NIV, up to 28 days
Nurse assessement of dyspnea during each NIV period measured by Likert scale (score range1-5; higher values represent a worst outcome) | after 1 hour of NIV, up to 28 days
Respiratory rate during SB periods | after 2 hours of SB in the 48 first hours, and every 4 hours thereafter, up to 28 days
Respiratory rate during NIV periods | after 1 hour of NIV, up to 28 days
Proportion of patients using accessory muscles during NIV periods | after 1 hour of NIV, up to 28 days
Daily arterial blood gases (ABG) (in terms of pH, PaCO2 and PaO2 measured between 8-10 am). | up to 28 days post-randomisation
Proportion of patients with premature NIV cessation (intolerance) (defined by agitation and/or mask removal, and/or patient's wish to interrupt session before) | 28 days post-randomisation
Proportion of patients refusing to resume NIV (despite meeting criteria) | 28 days post-randomisation
Proportion of patients who need secondary intubation and IMV | 28 days post-randomisation
Proportion of patients with nasal bridge ulceration | After 2 hours of SB in the 48 first hours, and every 4 hours thereafter; and after 1 hour of NIV; up to 28 days
Proportion of patients with eye irritation | After 2 hours of SB in the 48 first hours, and every 4 hours thereafter; and after 1 hour of NIV; up to 28 days
Proportion of patients with nasal congestion | After 2 hours of SB in the 48 first hours, and every 4 hours thereafter; and after 1 hour of NIV; up to 28 days
Proportion of patients with nasal/oral dryness | After 2 hours of SB in the 48 first hours, and every 4 hours thereafter; and after 1 hour of NIV; up to 28 days
Proportion of patients with gastric distension | After 2 hours of SB in the 48 first hours, and every 4 hours thereafter; and after 1 hour of NIV; up to 28 days
Proportion of patients with nosocomial pneumonia | After 2 hours of SB in the 48 first hours, and every 4 hours thereafter; and after 1 hour of NIV; up to 28 days
Proportion of patients with pneumothorax | After 2 hours of SB in the 48 first hours, and every 4 hours thereafter; and after 1 hour of NIV; up to 28 days
Proportion of patients with arterial hypotension | After 2 hours of SB in the 48 first hours, and every 4 hours thereafter; and after 1 hour of NIV; up to 28 days
Proportion of patients with nostril ulceration (including nasolabial angle, columella, nostril sill) | After 2 hours of SB in the 48 first hours, and every 4 hours thereafter; and after 1 hour of NIV; up to 28 days
Proportion of patients with nose bleeding | After 2 hours of SB in the 48 first hours, and every 4 hours thereafter; and after 1 hour of NIV; up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Damien Ricard, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Réanimation Médico-Chirurgicale, Hôpital Louis Mourier, Colombes, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ricard JD, Dib F, Esposito-Farese M, Messika J, Girault C; REVA network. Comparison of high flow nasal cannula oxygen and conventional oxygen therapy on ventilatory support duration during acute-on-chronic respiratory failure: study protocol of a multicentre, randomised, controlled trial. The 'HIGH-FLOW ACRF' study. BMJ Open. 2018 Sep 19;8(9):e022983. doi: 10.1136/bmjopen-2018-022983. PMID 30232113